CLINICAL TRIAL: NCT01732419
Title: Effects of Homebased Training With Telemonitoring Guidance in Low to Moderate Risk Patients Entering Cardiac Rehabilitation
Brief Title: Homebased Training With Telemonitoring Guidance in Low to Moderate Risk Patients Entering Cardiac Rehabilitation
Acronym: FIT@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, H.Kemps, MD, PhD, Maxima Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARDSS FIT@Home
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: Rehabilitation, exercise therapy, coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-based training (Experimental): After the first three supervised training sessions in the hospitals, patients in the home-based training group are instructed to wear a heart rate monitor during exercise training at home. Prescribed exercise exists of two or three exercise sessions per week, of one hour at 70 - 85% of their maximum heart rate.
  Once a week the heart rate data is uploaded and evaluated by an exercise specialist together with the patient by telephone.
  Interventions: Behavioral: Home-based training
- Centre-based training (Active Comparator): Patients in the centre-based training group will perform all trainings sessions under direct supervision of a physical therapist specialized in CR. Training sessions will be performed on an cycle ergometer, starting with a warm up phase of 5 min, followed by 50 min of cycling at 70-85% of the maximal HR and a cooling down period of 5 min. During the training period, physical therapists will record attendance, training duration and actual training intensity. After the 12-week training period patients receive individual advice from their physical therapist on physical activities.
  Interventions: Behavioral: Centre-based training

INTERVENTIONS:
Behavioral: Home-based training — Home-based exercise training for cardiac patients.
  Other Names: Homebased exercise training; Home-based cardiac rehabilitation
  Arms: Home-based training
Behavioral: Centre-based training — Usual exercise training in an outpatient setting.
  Other Names: Hospital-based training; Outpatient exercise training; Centre-based cardiac rehabilitation; hospital-based cardiac rehabilitation
  Arms: Centre-based training

SUMMARY:
Physical exercise training appears effective for low to moderate patients assigned to cardiac rehabilitation. However, adherence to cardiac rehabilitation is low and physical activity levels often drop after attending the last supervised rehabilitation session.

This study will compare home based physical exercise training including telemonitoring with regular centre based physical exercise training. Main outcome measures are the change in physical activity and the change in physical fitness (peak Oxygen uptake) after the initial rehabilitation period (12 weeks) and after 1 year. Secondary outcome measures are cost-effectiveness, training adherence, health-related quality of life and patient satisfaction.

DETAILED DESCRIPTION:
Physical training has beneficial effects on exercise capacity, cardiac function, quality of life and mortality in patients with acute cardiovascular syndrome or after cardiac surgery and is therefore one of the main aspects of cardiac rehabilitation. However, adherence to this therapy is low and effects tempt to decrease directly after the treatment period.

The objective of this study is to compare the effects of home-based exercise training (HT) with telemonitoring guidance and regular centre-based exercise training (CT) on physical fitness (PF), assessed by peak oxygen uptake, and physical activity (PA), assessed by physical activity energy expenditure (PAEE), in low to moderate risk cardiac rehabilitation (CR) patients. Secondary endpoints are cost-effectiveness, training adherence, health-related quality of life (QoL) and patient satisfaction.

Single-centre randomized controlled trial. CR patients are randomized to HT (n=45) or CT (n=45). Assessments are performed at baseline, 12 weeks and 1 year, consisting of maximal exercise testing with respiratory gas exchange analysis, assessment of PAEE, QoL (also at 6 months), patient satisfaction (at 12 weeks only) and health care costs (12 weeks, 6 months and 1 year) Study population: Low to moderate risk patients entering outpatient CR after an acute coronary syndrome or revascularization with internet access and PC at home.

12-week training program (24-36 one-hour sessions) at 70-85% of their maximal heart rate (HR). In the CT group training is supervised by a physical therapist; in the HT group training is performed in the home environment using a HR monitor to determine training intensity and with weekly feedback / motivation by an exercise specialist who has access to the online HR-data. After 12 weeks, subjects in the HT group are encouraged to continue using the HR monitor.

Main study parameters/endpoints: Primary endpoints: PF (peak oxygen uptake) and PA (physical activity energy expenditure, PAEE) assessed by a tri-axial accelerometer and HR monitor. Secondary endpoints: training adherence, QoL (SF-36) and patient satisfaction (CQ index).

Exercise training performed by patients after Acute Coronary Disease (ACS) and revascularization, classified as low to moderate risk, is considered to be safe. The training program that will be used in this study has been evaluated in a similar population of elderly cardiac patients without any documented harmful effects. In order to reduce potential risks of exercise training all patients perform a maximal cardiopulmonary exercise test at baseline, excluding patients with myocardial ischaemia and ventricular arrhythmias during exercise. The first three training sessions will be under supervision of trained physiotherapist in a clinical setting. The patients will receive a heart rate monitor and accelerometer to use at home. These monitors are developed and optimized to cause minimal physical discomfort and are non-invasive. During the measurement periods, all patients are asked to wear the monitors continuously for 5 days and to note the physical activities performed. The HT group will use the HR monitors during their physical trainings as well.

ELIGIBILITY:
Inclusion criteria:

* Patients with an ACS (including non ST and ST elevation myocardial infarction and unstable angina) or a cardiac revascularization procedure (PCI or CABG) entering outpatient CR at Maxima Medical Center.
* Indication for exercise training according to the Dutch clinical algorithm for assessment of patient needs in cardiac rehabilitation.
* Internet access and PC at home (i.e. more than 90 percent of the Dutch household)

Exclusion criteria:

* High risk according to the Dutch CR practice guideline.
* Systolic heart failure (left ventricular ejection fraction of more than 40 percent.
* New York Heart Association class III-IV (i.e. breathlessness during light exercise or at rest).
* Severe arrhythmia.
* Hemodynamically significant valvular disease.
* Implantable cardioverter-defibrillator (ICD) implantation
* Heart transplantation.
* Chronic angina or silent ischemia.
* Comorbidity impairing exercise capacity (e.g. COPD, diabetes mellitus, peripheral vascular disease and orthopedic or neurological conditions).
* Severe psychological or cognitive impairments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hareld Kemps, Dhr. MD., Principal Investigator — Maxima Medical Center
Locations (1):
- Máxima Medisch Centrum, Veldhoven, Netherlands

REFERENCES:
- [Derived] Kraal JJ, Peek N, Van den Akker-Van Marle ME, Kemps HM. Effects of home-based training with telemonitoring guidance in low to moderate risk patients entering cardiac rehabilitation: short-term results of the FIT@Home study. Eur J Prev Cardiol. 2014 Nov;21(2 Suppl):26-31. doi: 10.1177/2047487314552606. PMID 25354951
- [Derived] Kraal JJ, Peek N, van den Akker-Van Marle ME, Kemps HM. Effects and costs of home-based training with telemonitoring guidance in low to moderate risk patients entering cardiac rehabilitation: The FIT@Home study. BMC Cardiovasc Disord. 2013 Oct 8;13:82. doi: 10.1186/1471-2261-13-82. PMID 24103384

RESULTS

PARTICIPANT FLOW:
Groups:
- Home-based Training: After the first three supervised training sessions in the hospitals, patients in the home-based training group are instructed to wear a heart rate monitor during exercise training at home. Prescribed exercise exists of two or three exercise sessions per week, of one hour at 70 - 85% of their maximum heart rate.
  Once a week the heart rate data is uploaded and evaluated by an exercise specialist together with the patient by telephone.
  Home-based training: Home-based exercise training for cardiac patients.
Period: Overall Study
Arm/Group | Home-based Training | Centre-based Training
Started | 45 | 45
Completed | 37 | 41
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Population: Baseline measurements
Groups:
- Total: Total of all reporting groups
Arm/Group | Home-based Training | Centre-based Training | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (8.8) | 57.7 (8.7) | 59.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 40 | 40 | 80
Region of Enrollment [Number; unit: participants]
  Netherlands | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Physical Fitness
Description: Changes in peak oxygen uptake (VO2max) in mL O2/kg/min
Time Frame: Measured after 12 weeks and after one year
Population: patients finished the study
Measure: Mean (Standard Deviation); unit: ml O2/kg/min
Arm/Group | Home-based Training | Centre-based Training
Number analyzed (Participants) | 37 | 41
ml O2/kg/min
  Baseline | 24.4 (6.7) | 24.0 (5.6)
  Discharge CR (12 weeks) | 27.9 (7.5) | 26.5 (7.1)
  Follow up (1 year) | 27.7 (6.9) | 27.5 (8.1)

2. Primary Outcome: Physical Activity Level (PAL)
Description: PAL is calculated by combining data from an accelerometer with data from a heart monitor, after wearing both for five days continuously. To determine PAL, physical activity energy expenditure is divided by resting metabolic rate, calculated by the Harris-Benedict equation. PAL expressed a person's daily energy expenditure. When PAL is used to classify the intensity of an activity, PAL<3, PAL<6 and PAL>6 are characterized as light, moderate and vigorous intensity activities respectively. An average daily PAL of 1.2 represents the activity level of a bed-bound subject, while the average PAL for the adult population is 1.7.
Time Frame: measured after 12 weeks and after one year
Population: Patients finished the study
Measure: Mean (Standard Deviation); unit: PAL
Arm/Group | Home-based Training | Centre-based Training
Number analyzed (Participants) | 37 | 41
PAL
  Baseline | 2.09 (0.92) | 1.95 (0.86)
  Discharge CR (12 weeks) | 2.22 (0.99) | 2.38 (1.02)
  Follow up (1 year) | 2.14 (1.06) | 2.13 (1)

3. Secondary Outcome: Training Adherence
Description: Provides information on the average amount of training sessions were performed during the 12 week cardiac rehabilitation program. Both groups received the advice to train at least 2 times a week for 12 weeks (thus 24 sessions).
Time Frame: 12 weeks
Population: Patients finished the CR program
Measure: Mean (Standard Deviation); unit: Exercise sessions completed
Arm/Group | Home-based Training | Centre-based Training
Number analyzed (Participants) | 40 | 37
Exercise sessions completed | 22.0 (6.8) | 20.6 (4.3)

4. Secondary Outcome: Health Related Quality of Life
Description: Health-related quality of life will be assessed by the MacNew questionnaire. The items and scale are scored from 1 (low health-related Quality of Life) to 7 (High health-related Quality of Life).
Time Frame: measured at baseline, at discharge (12 weeks), and follow-up (one year)
Population: Patients finished the study
Measure: Mean (Standard Deviation); unit: Units of a scale
Arm/Group | Home-based Training | Centre-based Training
Number analyzed (Participants) | 37 | 41
Units of a scale
  Baseline | 5.62 (0.20) | 5.45 (0.14)
  Discharge CR (12 weeks) | 6.00 (0.13) | 5.90 (0.13)
  Follow up (one year) | 5.75 (0.10) | 5.43 (0.12)

5. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction is measured directly after CR discharge (12 weeks) using the Consumer Quality Index, a standardized survey method combining the inventory of patient experiences with an assessment of their priority. Results are provided on a scale of 1 (very low satisfaction) to 10 (very high satisfaction).
Time Frame: Measured at CR discharge (12 weeks)
Population: Patients finished the CR program (12 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Home-based Training | Centre-based Training
Number analyzed (Participants) | 40 | 43
units on a scale | 8.7 (1.0) | 8.1 (1.2)

ADVERSE EVENTS:
Time Frame: During the study period (1 year)
Description: The definition of adverse events did not differ from the clinicaltrials.gov definition.
Arm/Group | Home-based Training | Centre-based Training
Serious Adverse Events (participants affected / at risk) | 3/45 | 9/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home-based Training (N=45) | Centre-based Training (N=45)
Death (Vascular disorders) | 1 (1) | 0 (0)
Heart attack (Cardiac disorders) | 0 (0) | 1 (1)
Rehospitalization due to cardiac reasons (Cardiac disorders) | 2 (2) | 8 (8)

LIMITATIONS AND CAVEATS:
blinding of patients due to nature of the study protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No